CLINICAL TRIAL: NCT03789643
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of JTT-251 Administered for 24 Weeks to Participants With Pulmonary Arterial Hypertension (RELIEF-PAH)
Brief Title: Study to Evaluate Efficacy and Safety of JTT-251 in Participants With Pulmonary Arterial Hypertension
Acronym: RELIEF-PAH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Corporate decision, priority change
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT251-G-17-006
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: JTT-251; Pulmonary arterial hypertension; RELIEF-PAH; Six-minute walk distance (6MWD)
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- JTT-251 Dose 1 (Experimental): One dose of study drug by mouth daily for 24 weeks
  Interventions: Drug: JTT-251
- JTT-251 Dose 2 (Experimental): One dose of study drug by mouth daily for 24 weeks
  Interventions: Drug: JTT-251
- JTT-251 Dose 3 (Experimental): One dose of study drug by mouth daily for 24 weeks
  Interventions: Drug: JTT-251
- Placebo (Placebo Comparator): One dose of study drug by mouth daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JTT-251 — Active drug tablets containing JTT-251
  Arms: JTT-251 Dose 1; JTT-251 Dose 2; JTT-251 Dose 3
Drug: Placebo — Placebo tablets matching in appearance to the active drug tablets
  Arms: Placebo

SUMMARY:
Study to evaluate the efficacy, safety, tolerability and pharmacokinetics of JTT-251 administered for 24 weeks in participants with pulmonary arterial hypertension (PAH)

DETAILED DESCRIPTION:
This is a study to evaluate the efficacy, safety, tolerability and pharmacokinetics of JTT-251 administered for 24 weeks in participants with pulmonary arterial hypertension (PAH). Participants completing this study (RELIEF-PAH) will be eligible to enroll in an open-label extension study (RELIEF-PAH OLE) to evaluate the long-term efficacy, safety, tolerability and pharmacokinetics of JTT-251 in participants with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAH as classified by idiopathic, heritable, drug and toxin- induced, congenital heart disease or associated with connective tissue disease (i.e., WHO Group 1)
* Clinical diagnosis of PAH confirmed by RHC at any time prior to Visit 1
* WHO functional status of Class II-IV at Visit 1
* Two 6MWD test measurements between 100 and 450 meters with a relative difference of ≤15%. The baseline 6MWD test must be performed at Visit 2 before randomization.
* Have a qualifying RHC performed between Visit 1 and Visit 2
* On stable dose(s) of guideline-directed medical therapy for PAH (endothelin receptor antagonists, phosphodiesterase type-5 (PDE-5) inhibitors, soluble guanylate cyclase stimulators and prostacyclin pathway analogs) for at least 90 days prior to the qualifying RHC

Exclusion Criteria:

* PAH associated with portal hypertension, human immunodeficiency virus (HIV), schistosomiasis or sickle cell disease as well as participants with pulmonary parenchymal disease or thromboembolic disease
* Known significant left heart disease including: left ventricular dysfunction (i.e., left ventricular ejection fraction <35%); hemodynamically compromising, symptomatic, or severe aortic stenosis, aortic regurgitation, mitral stenosis, mitral regurgitation
* Pulmonary hypertension belonging to WHO groups 2 to 5
* Moderate to severe obstructive lung disease defined as forced expiratory volume in 1 second (FEV1) <55% of predicted value
* Moderate to severe restrictive lung disease defined as total lung capacity (TLC) <60% of predicted value
* Acute decompensated heart failure or hospital admission for worsening PAH symptoms within 30 days prior to the qualifying RHC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in six-minute walk distance (6MWD) compared to baseline | 24 Weeks
Change in World Health Organization (WHO) functional classification compared to baseline | 24 Weeks
Change in pulmonary vascular resistance (PVR) compared to baseline | 4, 12, 24 and 28 Weeks
  Assessed by right heart catheterization (RHC)

SECONDARY OUTCOMES:
Number of adverse events | 28 Weeks
JTT-251 trough plasma concentrations | 4, 12 and 24 Weeks

IPD SHARING:
Plan to Share IPD: No